CLINICAL TRIAL: NCT05479292
Title: Medical Care of Cancer Patients During the COVID-19 Pandemic - an Analysis of Health Insurance Claims Data
Brief Title: Allocating Resources for Cancer Care in Times of the Sars-CoV-2 Outbreak. Health Care Research
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); AOK PLUS (Industry); Medizinische Fakultät der Martin-Luther-Universität Halle-Wittenberg (Unknown); Ruhr-Universität Bochum (Unknown)
Responsible Party: Sponsor
Other Study IDs: CancerCOVID-HCR
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer (CRC) and Pancreatic Cancer (PaCa)
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sars-CoV-2 outbreak — Sars-CoV-2 pandemic's impact on provision of healthcare for cancer patients

SUMMARY:
The focus on treatment of COVID19 patients during the Sars-CoV-2 outbreak has most likely implications for the extent and quality of diagnosis and treatment of non-COVID19 patients. Medical care of cancer patients is a particularly sensitive area. To draw holistic conclusions, it is necessary to analyze the provision of healthcare as broadly as possible with regard to the dimensions of access, processes and outcome during the Sars-CoV-2 pandemic. This will be implemented exemplarily for the early detection, diagnosis and treatment of colorectal cancer (CRC) and pancreatic cancer (PaCa) in Saxony. Patients with diagnosis, treatment or early detection measures for type 2 diabetes (T2D), coronary heart disease (CHD) and multiple sclerosis (MS) serve as comparison groups.

DETAILED DESCRIPTION:
For a realistic assessment, the situation will be compared with the situation before the Sars-CoV-2 pandemic while considering confounders and effect modifiers. The evaluation is based on pseudonymised routine statutory health insurance (SHI) data of the AOK PLUS for Saxony.

As data sources, SHI data of the AOK PLUS Saxony for the period 2015 to 4th quarter 2020 and publicly available data on COVID19 are used. The differentiation between incidence and prevalent diseases is based on a 4-year washout period, so that the health care situation can be compared between 2019 (pre-period) and 2020 (post-period). Patients with confirmed diagnoses of CRC and PaCa or early detection measures regarding CRC are investigated. These will be contrasted to patients with confirmed diagnoses of T2D, CHD, and MS or early detection measures regarding T2D.

The differentiation of subgroups as confounders or effect modifiers is taken into account. Subgroups are considered with respect to the factors age groups, gender, Elixhauser comorbidities, metastasis y/n, residential regions (postal code 3 digits), characteristics of the treating institution and possibly seasonal effects.

Aims:

Analysis of the differences in the health care provision situation during the Sars-CoV-2 outbreak compared to the time before.

Research questions:

1. (How) did the situation of health care for cancer patients change due to the outbreak of Sars-CoV-2? Which changes could be observed in the dimensions access to care, quality or guideline adherence in medical care and outcome?
2. Did the focus on COVID19 patients have an impact on the diagnosis or early detection of cancer in Saxony?
3. Are the observed effects differential with respect to the diseases, especially when comparing CRC and PaCa with the control group regarding T2D and CHD?

ELIGIBILITY:
Inclusion Criteria:

* Resident of Saxony, Germany with health insurance coverage provided by AOK PLUS
* Diagnosis of colorectal cancer, pancreatic cancer, type 2 diabetes, coronary heart disease or multiple sclerosis between in 2019 or 2020 according to ICD-10

Exclusion Criteria:

* Change of health insurance provider between 2015 and 2020
* Born after 2014
* Deceased between 2015-2018

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Saxony, Germany with continuous health insurance coverage provided by the AOK PLUS from 2015 - 2020 with a diagnosis of colorectal cancer, pancreatic cancer, type 2 diabetes, coronary heart disease or multiple sclerosis in 2019 or 2020 according to ICD-10
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of confirmed diagnoses (new cases of CRC or PaCa) | Comparison of 2019 to 2020
Number of colonoscopies | Comparison of 2019 to 2020

SECONDARY OUTCOMES:
Number of hospitalizations | Comparison of 2019 to 2020
Number of surgeries/systemic therapies related to cancer after onset of disease | Comparison of 2019 to 2020

OTHER OUTCOMES:
Pathway of health care | Comparison of 2019 to 2020

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schmitt, Dr. med., Principal Investigator — Technische Universität Dresden
Locations (1):
- ZEGV, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No